CLINICAL TRIAL: NCT00723580
Title: Actigraphic Analysis of Treatment Response in a Six Year Old Girl With Kabuki Syndrome
Brief Title: Actigraphic Analysis of Treatment Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Child Psychopharmacology Institute (Other)
Responsible Party: Principal Investigator, Bill J. Duke, M.A., Ph.D., ABMPP, Director, Child Psychopharmacology Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Act1
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Results first posted 2010-12-14 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-07

CONDITIONS: Sleep Disorders, Circadian Rhythm; Insomnia; Psychomotor Agitation
Keywords: Kabuki Syndrome; Actigraphy; Treatment Response Measurement
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Sleep Initiation and Maintenance Disorders; Psychomotor Agitation; Kabuki syndrome | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sleep and Activity by Treatment Condition (Experimental): Actigraphic measurements were obtained by attaching an actigraphic watch device to the child's non-dominant wrist. The measurements will include three separate three week periods beginning with a baseline period and the period in which the child's pharmacological treatment was initiated. Two additional three week actigraphic measurement periods will occur at 22 months post-baseline period and at 23 months post-baseline period. The resulting five treatment conditions were: 1. Baseline no medication 2. Risperidone .25 mg at bedtime (q.h.s.) x 7 days 3. Risperidone .25 mg twice daily (b.i.d.) 4. Risperidone .25 mg three times a day (t.i.d.) and 5. Risperidone .5 mg three times a day (t.i.d.). Sleep and activity will be evaluated by treatment conditions.
  Interventions: Drug: risperidone

INTERVENTIONS:
Drug: risperidone — Five treatment conditions: 1. Baseline no medication 2. Risperidone .25 mg at bedtime (q.h.s.) x 7 days 3. Risperidone .25 mg twice daily (b.i.d.) 4. Risperidone .25 mg three times a day (t.i.d.) and 5. Risperidone .5 mg three times a day (t.i.d.).
  Other Names: Actigraphic measurements

SUMMARY:
The study examines and illustrates the utility of utilizing actigraphic measurements to assess treatment response.

DETAILED DESCRIPTION:
Actigraphic measurements will be recorded every 30 seconds and will be recorded for an 11 day baseline period, followed by a 10 day period of the initial pharmacological interventions. The non-invasive nature of watch-like actigraphy devices is particularly attractive for use in pediatric populations. Meaningful treatment response measurements are obtained when actigraphic data is combined with psychometric and observational repeated measurements. Subsequent to the initial data collection the parent consented and the child assented to extend the study and continue measurements.

The case study included baseline and repeated psychological, observational and actigraphic measurements that were initiated prior to treatment with risperidone and repeated throughout the treatment process with the final data collected in July 2010.

The Personality Inventory for Children (PIC) is an objective multidimensional measurement of affect, behavior, ability and family function. The PIC was administered prior to treatment with risperidone and repeated after 22 months of treatment. The PIC serves as both an actuarial pre-treatment diagnostic tool as well as a post-treatment repeated measurement indicating treatment associated change.

A primary observer (mother) was trained to report symptom percentages present since previous observations utilizing the operationally defined and observer defined items of the systematic observation scale throughout the treatment process.

Actigraphic measurements provide a basis by which to measure sleep and sleep onset latency as well as periods of mobility and immobility. When programmed to record activity every thirty seconds, thousands of measurements are quickly captured.

Actigraphic measurements were made utilizing a watch-like actigraphic device with an 11 day baseline actigraphic measurement period and continued measurements that included the initiation of a Once-Daily, Bedtime (q.h.s.) pharmacological intervention for 6 days, followed by a planned adjustment to Twice a Day (b.i.d.) dosing that was measured for an additional 4 days. Repeated actigraphic studies were subsequently conducted after 22 months of risperidone treatment and were collected along with the repeated observational and psychometric data.

This case study explores activity and sleep characteristics related to behavioral characteristics and treatment response and the utility of single subject repeated actigraphic, psychometric and observational measurements and monitoring of treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Kabuki Syndrome
* Medication Naive
* Single subject preparing to receive pharmacological intervention

Exclusion Criteria:

* Inability to wear actigraphy device

Ages: 2 Years to 10 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2008-05; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bill J Duke, M.A., Ph.D., Principal Investigator — Child Psychopharmacology Institute
Locations (1):
- Child Psychopharmacology Institute, Fargo, North Dakota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A six year old child with Autism Spectrum Disorder (pervasive developmental disorder) and Kabuki Syndrome anticipating a pharmacological intervention was evaluated for sleep and behavioral disturbances. She was invited to participate, her parents provided consent and the child acknowledged her assent.
Pre-assignment Details: The child had previously not responded to multiple medication trials, was stimulated by diphenylhydramine, over-sedated on clonidine and had mood destabilization when tried on mirtazapine. The child received no medication for the month preceding the initiation of the study.
Groups:
- Actigraphic (Activity Count) Measurement of Sleep and Activity: Actigraphic measurements obtained by attaching an actigraphic watch device to the child's non-dominant wrist obtain measurements that occur every thirty seconds for a duration of approximately 21 days. These measurements reflect treatment condition sleep characteristics where sleep is indicated by activity counts below 40. Three 21 day actigraphic measurement periods occurred with the initial measurement occurring through baseline period and the period in which the child's pharmacological treatment was initiated. The second and third, 21 day periods of Actigraphic measurement occurred at 22 and 23 months from baseline. Five treatment conditions during the measurement periods including 1. baseline no medication 2. risperidone .25 mg at bedtime for 7 days (q.h.s.) 3. risperidone twice daily (b.i.d.) 4. risperidone .25 mg three times a day (t.i.d.) and 5. risperidone .50 mg three times a day (t.i.d.)
Period: Overall Study
Arm/Group | Actigraphic (Activity Count) Measurement of Sleep and Activity
Started | 1 (Study was extended with continued repeated measurements.)
Baseline Measurements | 1 (Actigraphic, Psychometric and Observational Baseline Data Collected.)
Completed | 1 (Completion of repeated Measurements)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Actigraphic (Activity Count) Measurement of Sleep and Activity
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Actigraphic Measurement of Treatment Conditions
Description: The child's impulsivity and inability to sleep represented a significant symptom and risk factor. Impulsivity and sleep will be actigraphically assessed by treatment conditions.
Time Frame: May 12- July 14, 2010
Population: Single subject repeated Actigraphic(at thirty second intervals), observational (every two months) and psychometric (baseline and at 23 months) measurements of a child anticipating pharmacological treatment. Actigraphic measurements (three 21 day periods) over five treatment conditions that included a non-medication baseline and spanned 23 months.
Measure: Mean (Standard Deviation); unit: activity
Units Other Than Participants: Activity counts
Arm/Group | Actigraphic (Activity Count) Measurement of Sleep and Activity
Number analyzed (Participants) | 1
Number analyzed (Activity counts) | 191235
activity
  Baseline No Medication Midnight to 1:00 AM | 55.02 (206.432)
  risperidone .5 mg t.i.d. Midnight to 1:00 AM | 9.94 (51.651)

2. Secondary Outcome: Systematic Observation Scale Item: Percentage of Impulsivity Observed
Description: The Systematic Observation Scale utilizes single-subject repeated measurements. Symptoms and issues of interest are defined and a variety of frequency and sampling methods can be applied. The Systematic Observation Scale was designed so Primary Observers (parents, guardians, self observers or others) can make pre-treatment and subsequent observations to track, document and evaluate symptom variation over the course of an illness. The measurement utilized is the percentage of time the symptom is observed by the primary observer since the previous observation.
Time Frame: May-7-2008 to July -14-2010
Reporting Status: Not Posted

3. Secondary Outcome: Systematic Observation Scale: Percentage of Irritability Observed
Time Frame: May-7-2008 to July -14-2010
Reporting Status: Not Posted

4. Secondary Outcome: Systematic Observation Scale: Percentage of Distractibility Observed
Time Frame: May-7-2008 to July -14-2010
Reporting Status: Not Posted

5. Secondary Outcome: Systematic Observation Scale: Percentage of Hyperactivity Observed
Time Frame: May-7-2008 to July -14-2010
Reporting Status: Not Posted

6. Secondary Outcome: The Personality Inventory for Children: Adjustment Scale
Description: This scale measures general personality adjustment reflecting a dimension associated with highly adaptive to maladaptive adjustment. The Personality Inventory for Children (PIC) is an age and gender referenced objective multidimensional measurement of affect, behavior, ability and family function. The PIC was administered prior to treatment with risperidone and repeated after 22 months of treatment. The PIC serves as both an actuarial pre-treatment diagnostic tool as well as a post-treatment repeated measurement indicating treatment and developmentally associated change.
Time Frame: May-7-2008 to July -14-2010
Reporting Status: Not Posted

7. Secondary Outcome: The Personality Inventory for Children: Achievement Scale
Description: The factors that underlie this scale are academic ability, poor achievement, impulsivity, limited concentration and over or under-assertiveness with peers. The Personality Inventory for Children (PIC) is an age and gender referenced objective multidimensional measurement of affect, behavior, ability and family function.
Time Frame: May-7-2008 to July -14-2010
Reporting Status: Not Posted

8. Secondary Outcome: The Personality Inventory for Children: Somatic-Physiological Scale
Description: The factors that underlie this scale are fatigue, aches and pains, insomnia, somatic response to stress and malingering. The Personality Inventory for Children (PIC) is an age and gender referenced objective multidimensional measurement of affect, behavior, ability and family function.
Time Frame: May-7-2008 to July -14-2010
Reporting Status: Not Posted

9. Secondary Outcome: The Personality Inventory for Children: Delinquency Scale
Description: The factors that underlie this scale are poor frustration tolerance, irritability, sadness, lack of interest, hostility,limited social participation and resistance to authority. The Personality Inventory for Children (PIC) is an age and gender referenced objective multidimensional measurement of affect, behavior, ability and family function.
Time Frame: May 7, 2008-July 14,2010
Reporting Status: Not Posted

10. Secondary Outcome: The Personality Inventory for Children: Withdrawal Scale
Description: The factors that underlie this scale are physical isolation, Shyness, isolation from peers, emotional distance and isolated intellectual interests. The Personality Inventory for Children (PIC) is an age and gender referenced objective multidimensional measurement of affect, behavior, ability and family function
Time Frame: May-7-2008 to July -14-2010
Reporting Status: Not Posted

11. Secondary Outcome: The Personality Inventory for Children: Social Skills Scale
Description: The factors that underlie this scale are social success, social rejection, adults as only social contacts, and the ability to lead and follow. The Personality Inventory for Children (PIC) is an age and gender referenced objective multidimensional measurement of affect, behavior, ability and family function.
Time Frame: May-7-2008 to July -14-2010
Reporting Status: Not Posted

12. Secondary Outcome: The Personality Inventory for Children: Family Relations Scale
Description: The factors that underlie this scale are family stability, inter-parent communication, presence of love and happiness in the home and appropriateness of discipline. The Personality Inventory for Children (PIC) is an age and gender referenced objective multidimensional measurement of affect, behavior, ability and family function.
Time Frame: May-7-2008 to July -14-2010
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 23 months
Description: Treatment monitoring was occurring throughout the study
Arm/Group | Actigraphic (Activity Count) Measurement of Sleep and Activity
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
This single case study has limited generalizability in that these results may not apply to others. The methods explored, however, may apply to others and Single-subject repeated measurements can provide valuable clinical and scientific data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes